CLINICAL TRIAL: NCT01538108
Title: The Use of NMB Drug Ejecting Balloon for Arteriovenous (AV) Dialysis Fistulae
Brief Title: Study of NMB (Company's Name) Drug Ejecting Balloon for Arteriovenous Fistulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: N.M.B. Medical Applications Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMB AVS P
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Obstructive Lesions of Arteriovenous Dialysis Fistulae

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- NMB's PTA Balloon catheter with paclitaxel (Experimental)
  Interventions: Device: PTA Balloon catheter with paclitaxel
- Standard Angioplasty Balloon (Active Comparator)
  Interventions: Procedure: Plain Balloon angioplasty (PBA)

INTERVENTIONS:
Device: PTA Balloon catheter with paclitaxel — patients treated by the NMB's PTA Balloon catheter with paclitaxel
  Arms: NMB's PTA Balloon catheter with paclitaxel
Procedure: Plain Balloon angioplasty (PBA) — PBA
  Arms: Standard Angioplasty Balloon

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the use of NMB's percutaneous transluminal angioplasty (PTA) Balloon.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years and older
* Patients with arteriovenous fistula with obstructive lesion
* Patient who is willing and able to sign a written informed consent

Exclusion Criteria:

* age < 18
* female with child bearing potential
* Previous participation in another study with any investigational drug or device within the past 30 days
* Life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Restenosis Rate | 6 months

SECONDARY OUTCOMES:
Restenosis rate | 1,3 and 12 months
Easy insertion and removal | intraprocedural
Major adverse events | intraprocedural, 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel